CLINICAL TRIAL: NCT03703284
Title: Molecular Mechanisms Underlying the Occurrence of Malignant Cerebral Edema After Large Hemispheric Infarction (LHI)
Brief Title: Molecular Mechanisms of Malignant Cerebral Edema After LHI
Acronym: LHI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yan Zhang, Associate Professor, Xuanwu Hospital, Beijing
Other Study IDs: LHI
Record Dates: First submitted 2018-09-05; First posted 2018-10-11 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Cerebral Edema
Keywords: mechanism,; cerebral edema,; large hemispheric infarction
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LHI Hernia: Acute (<=48h) large hemispheric infarction (LHI) patients who developed cerebral hernia in 5 days post-stroke
  Interventions: Other: Treatments to reduce intracranial pressure
- LHI Non-Hernia: Acute (<=48h) large hemispheric infarction (LHI) patients without cerebral hernia in 5 days post-stroke
  Interventions: Other: Treatments to reduce intracranial pressure
- Healthy control: Healthy individuals

INTERVENTIONS:
Other: Treatments to reduce intracranial pressure — Drugs such as mannitol, glycerin fructose, etc and/or surgery
  Groups: LHI Hernia; LHI Non-Hernia

SUMMARY:
The study is to explore the molecular mechanisms underlying the occurrence of malignant cerebral edema (cerebral hernia) after large hemispheric infarction. Acute LHI (<=48h) patients that develop cerebral hernia or not within 5 days post-stroke onset, as well as the healthy controls will be studied. The participants will be followed for up to 6 months post stroke-onset, and their modified Rankin Scale (mRS) will be recorded. A mRS score of 0-4 is considered as a favorable outcome while a score of 5-6 as an unfavorable one.

DETAILED DESCRIPTION:
A total of 80 patients with acute large hemispheric infarction (LHI) within 48h after occurrence admitted into NICU of Xuanwu Hospital as well as 40 healthy volunteers will be recruited. The patients' baseline characteristics, treatment and changes of clinical conditions will be recorded, and ICP monitoring (D2-D7 post-stroke), chest X-ray (D2, D7, D14 post-stroke), ECG (D2, D7, D14 post-stroke), cerebral vascular ultrasound, TCD and head MRI (T1WI, T2WI, FLAIR, DWI) on D2 and D14 post-stroke will be performed. Blood samples from both the LHI patients (D2, D4, D7, and D14 post-stroke) and the controls will be analyzed for NEU, TNF-alpha, IL-1b, IL-6, IL-8, IL-17, ICAM-1, VCAM-1, MPO, NE, MMP-9,miRNA, free dsDNA, H3CIT and NETosis levels. All patients were treated for brain edema with osmotic medications-either intravenous 20% mannitol or 10% hypertonic saline. In addition, some patients were treated with decompressive surgery.The patients will be followed up to 6 months and their modified Rankin Scale (mRS) will be recorded. A mRS score of 0-4 is considered as a favorable outcome while a score of 5-6 as an unfavorable one. Statistical differences in the different parameters between different groups at different time points will be analyzed by SPSS 22.0 software.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-80 years old;
* 2. Clinical diagnosis of large hemispheric infarction
* 3. Within 48h after stroke onset.

Exclusion Criteria:

* 1. Clinical diagnosis of severe infection;
* 2. Clinical diagnosis of severe heart, liver or kidney diseases;
* 3. Clinical diagnosis of bleeding tendency, active bleeding or hematological diseases;
* 4. Malignant tumor;
* 5. Modified Rankin Scale (mRS)<2 before stroke onset.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that are recruited into the Neuro-intensive care unit (NICU) of Xuanwu Hospital during 2018.1.1-2022.12.31
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 6 months after stroke onset
  modified Rankin Scale: 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead. A score of 0-4 is considered as a favorable outcome, whereas a score of 5-6 was considered as an unfavorable one. The reasons for death should be also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M.D., PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No